CLINICAL TRIAL: NCT05920395
Title: Mechanisms of Electroacupuncture for Functional Dyspepsia Based on "Enterotypes" and Metabolomics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WZ22A06
Record Dates: First submitted 2023-06-05; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; Electroacupuncture; Intestinal flora

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy control group (No Intervention): 26 healthy volunteers without any intervention, detecting gastrointestinal hormone levels and intestinal microbiota and their metabolites.
- PDS electroacupuncture group (Experimental): Each with 26 patients who were treated with electro-acupuncture.
  Interventions: Other: Electro-acupuncture
- PDS sham electroacupuncture group (Sham Comparator): Each with 26 patients. Shallow acupuncture needles are used and then disconnected from the electrode.
  Interventions: Other: Sham electro-acupuncture group
- EPS electroacupuncture group (Experimental): Each with 26 patients who were treated with electro-acupuncture.
  Interventions: Other: Electro-acupuncture
- EPS sham electroacupuncture group (Sham Comparator): Each with 26 patients. Shallow acupuncture needles are used and then disconnected from the electrode.
  Interventions: Other: Sham electro-acupuncture group

INTERVENTIONS:
Other: Electro-acupuncture — Patients lie supine on the treatment bed, and after routine disinfection, a 0.30×60mm or 0.30×40mm disposable sterile acupuncture needle is inserted directly into the acupoint. Once obtaining qi, the needle is manipulated with even reinforcing and reducing techniques to maintain needle sensation. Acupoints selected include Zhongwan, Zusanli, Neiguan, and Tianshu, connected to the 6805-All electro-acupuncture therapy device. Zhongtuo and Tianshu acupoints are connected to a set of electrodes, with the positive pole connected to Zhongtuo and the negative pole connected to one side of Tianshu. The stimulation uses sparse and dense wave pulses with a frequency of 2Hz/100Hz, with the stimulation intensity determined based on individual patient tolerance. Each session lasts for 30 minutes, with a treatment frequency of once every other day, for a total of 4 weeks.
  Arms: EPS electroacupuncture group; PDS electroacupuncture group
Other: Sham electro-acupuncture group — Shallow acupuncture needles are used and then disconnected from the electrode. They are tied with black tape and connected to the sham electrode. The device is not powered on, and the rest of the treatment is the same as the electro-acupuncture group.
  Arms: EPS sham electroacupuncture group; PDS sham electroacupuncture group

SUMMARY:
The goal of this clinical trial is to explore the clinical efficacy and possible mechanisms of electroacupuncture treatment for functional dyspepsia (FD). The main question it aims to answer are:

* Differences in the effects of electroacupuncture and sham electroacupuncture intervention on FD.
* Differences in gastrointestinal hormone levels and gut microbiota and their metabolites between healthy individuals and FD patients.

Participants receive electroacupuncture and sham electroacupuncture interventions respectively. Before and after the intervention, the clinical symptom score, gastrointestinal symptom evaluation scale, gastrointestinal symptom score questionnaire, and functional dyspepsia quality of life scale of the subjects will be observed. The levels of gastrointestinal hormones MTL, Ghrelin, 5-HT, CCK, PYY, and GLP-1 will be measured, as well as the changes in microbial diversity and SCFAs in their metabolites in feces, A follow-up visit will be conducted one month after the intervention for all participants.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is a common and difficult clinical disease, and there is currently no effective treatment plan. Electroacupuncture is commonly used in clinical practice, but there is a lack of high-quality clinical evidence of its effectiveness. This study explores the clinical efficacy and possible mechanisms of electroacupuncture in the treatment of FD.

The study set up a healthy control group and an FD group. The FD group was divided into PDS type and EPS type according to their classification, and received electroacupuncture and sham electroacupuncture intervention, respectively. Before and after intervention, the clinical symptom score, gastrointestinal symptom evaluation scale, gastrointestinal symptom score questionnaire, and functional dyspepsia quality of life scale of the participants were observed. The levels of gastrointestinal hormones MTL, Ghrelin, 5-HT, CCK, PYY, GLP-1 were measured, and changes in fecal microbiota diversity and SCFAs in their metabolites were also detected. A follow-up visit will be conducted one month after the intervention for all participants.

Experiment 1: Observing the differences in various indicators between healthy individuals and FD patients Grouping: ① Healthy control group: 26 healthy volunteers, without any intervention, were tested for gastrointestinal hormone levels, gut microbiota, and their metabolites.② FD group: A total of 104 patients were included, and the levels of gastrointestinal hormones, gut microbiota, and their metabolites were detected after inclusion. The differences in gut type between the two groups of patients were analyzed.

Experiment 2: Observing the Effect of Electroacupuncture on FD Patients Grouping: The 104 FD patients included as required included 52 PDS type and 52 EPS type. Both types of patients were randomly assigned to the electroacupuncture group and the sham electroacupuncture group, with 26 patients in each group. It is divided into PDS electroacupuncture group (Group A), PDS sham electroacupuncture group (Group B), EPS electroacupuncture group (Group C), and EPS sham electroacupuncture group (Group D).

① Electroacupuncture group: including Group A and Group C, with 26 cases each, all receiving electroacupuncture treatment. The patient lies on his back on the treatment bed. After routine disinfection, a 0.30X50mm or 0.30X40mm disposable sterile acupuncture and moxibustion needle is directly punctured into the acupoint. After getting qi, the needling sensation is maintained by the manipulation of leveling, reinforcing and reducing. Point selection: Zhongwan, Zusanli, Neiguan, and Tianshu, connected to the 6805-AII electroacupuncture treatment instrument; Connect one set of electrodes to Zhongwan and Tianshu acupoints, with the positive electrode connected to Zhongwan acupoint and the negative electrode connected to Tianshu acupoint on one side; Using dense wave pulse stimulation with a frequency of 2Hz/100Hz, with a stimulation intensity that the patient can tolerate, 30 minutes each time, treated once every other day for a total of 4 weeks.

② False electroacupuncture: including group B and group D, with 26 cases each, with shallow acupuncture. After disconnecting the end of the electrode and binding it with black tape, the false electrode was connected without being electrified, and the rest were the same as the electroacupuncture group.

The positioning of acupoints shall refer to the positioning standards in the new century national planning textbook for higher Chinese medicine colleges and universities, "Meridian and Acupoint Science," edited by Shen Xueyong. A follow-up visit will be conducted one month after the intervention for all subjects.

During the intervention, all subjects did not take drug treatment. If the corresponding symptoms of the subjects such as abdominal pain, abdominal burning, early satiety and so on were significantly aggravated, the subjects would be given symptomatic treatment of the emergency drug pantoprazole sodium enteric coated tablets when the investigator diagnosed that drug intervention was needed. Participants can also consider choosing to seek treatment at the gastroenterology outpatient department. If needed, they can assist in contacting a specialist to provide corresponding professional diagnosis and treatment advice. Subjects receiving emergency medication or other medications that affect gastrointestinal motility need to terminate the study. If they have completed 1/2 course of treatment, the corresponding outcome indicators should be included in the efficacy statistics.

ELIGIBILITY:
FD diagnostic criteria:

Functional dyspepsia diagnostic criteria: According to the Rome IV diagnostic criteria for functional dyspepsia (2016).

Symptoms:①Early satiety; ②Postprandial fullness and bloating; ③Epigastric pain;④ Epigastric burning.

One or more of these four symptoms must be met, and there must be no evidence of structural diseases (including gastroscopy, etc.) that can explain these symptoms. In addition, the detailed diagnostic criteria for postprandial distress syndrome (PDS) or epigastric pain syndrome (EPS) must also be met.

The diagnosis of EPS meets the following criteria.

1. Meeting at least one of the following criteria for at least one day per week.

   ① Postprandial fullness and bloating (of such a degree as to affect daily living);

   ② Early satiety (of such a degree as to result in inability to finish a normal meal).
2. Routine examinations (including gastroscopy) did not reveal any systematic, organic, or metabolic diseases that could explain the above symptoms;
3. Symptoms must have appeared for at least six months prior to diagnosis, and met the above criteria for the past three months.

The diagnostic criteria for EPS include meeting at least one of the following criteria for at least one day per week:

1. Epigastric pain (of such a degree as to affect daily living);
2. Epigastric burning (of such a degree as to affect daily living);
3. Routine examinations (including gastroscopy) did not reveal any systematic, organic, or metabolic diseases that could explain the above symptoms;
4. Symptoms must have appeared for at least six months prior to diagnosis, and met the above criteria for the past three months.

Inclusion criteria

1. Meeting the Western medicine diagnostic criteria for FD;
2. Aged 18-65 years (inclusive of 18 and 65 years old);
3. Not having taken any gastrointestinal prokinetic drugs for at least 15 days before treatment, and not having participated in any other clinical studies;
4. Voluntary signing of an informed consent form for this study. Note: Only patients who meet all four of the above criteria can be included in this study.

Exclusion criteria

1. Pregnant or lactating women;
2. Patients with severe organic digestive system diseases indicated by endoscopic examination, such as severe dysplasia or mucosal erosion, or pathological indication of malignancy;
3. Patients with endocrine, cardiovascular, cerebrovascular, hematopoietic system, or neurological diseases such as diabetes, severe coronary heart disease, hypoglycemia, or hemiplegia;
4. Patients with mental illness,infectious diseases, progressive malignant tumors,or life- threatening diseases;
5. Patients who are afraid of acupuncture, have allergies or are allergic to medical supplies.

Note: Patients who meet any of the above criteria will be excluded.

Removal criteria

1. Cases that are mistakenly included due to concealment of illness information or failure to meet inclusion criteria should be excluded;
2. Participants with poor compliance or those who withdraw from the study on their own during the treatment period, or those who use treatment methods prohibited by this protocol during the study phase;
3. Participants who experience severe adverse events or complications and are unable to continue the treatment, and the trial is terminated;
4. Participants who do not follow the prescribed treatment or whose data is incomplete, affecting efficacy and safety evaluation.

Dropout criteria Participants who have been included but are unable to participate in the trial on time, or who do not follow the trial requirements, or who drop out during treatment.

The handing of exclusion and dropout When a participant drops out, the researcher should contact them as much as possible through house visits, scheduled phone calls, letters, etc., to inquire about the reasons for dropout. record the date of the last treatment, and complete the evaluation items that can be completed. All cases of exclusion and dropout will be subjected to intention-to-treat analysis after the end of the trial.

Research Termination Criteria

1. If the condition worsens during the experiment or other serious illness occurs, it is determined that participation needs to be terminated or other treatments are necessary.
2. If a serious adverse event occurs during the experiment that prevents further participation.
3. The investigator should record the reason and time for withdrawing from the study. Those who have completed more than half of the treatment should be included in the efficacy statistics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall efficacy evaluation | up to 4 weeks
  Refer to the efficacy criteria in the "Draft of Integrated Traditional Chinese and Western Medicine Diagnosis and Treatment Plan for Functional Dyspepsia", and evaluate the efficacy based on four levels: clinical cure, marked improvement, improvement, and inefficacy. Calculate the efficacy index based on the total symptom score. Efficacy index = {(pre-treatment total symptom score - post-treatment total symptom score) ÷ pre-treatment total symptom score} × 100%.
  Clinical Cure: Efficacy Index > 85%; Marked Improvement: Efficacy Index 5%-85%; Improvement: Efficacy Index 26%-50%; Inefficacy: Efficacy Index < 26%.
Gastric electrogastrography (EGG) testing | baseline, pre-intervention
  The Hefei Scientific Experimental Instrument Factory's GAP-24A high-resolution gastrointestinal electrogastrography analysis system is used for testing. In the fasted state, the subject lies in a supine position, and electrodes are placed on the upper abdomen at the first lead of the gastric antrum (2-4 cm to the right of the midpoint between the xiphoid process and umbilicus) and the second lead of the gastric body (3-5 cm to the left of the midpoint between the xiphoid process and umbilicus, 1 cm upward). Conductive gel is applied locally to the skin, and a baseline EGG recording is made before conducting gastric EGG evaluation. After recording for 30 minutes, subjects are given a standard meal (50% carbohydrates, 25% protein, 25% fat, total energy intake of 570kcal, and 150mL water), which they eat within 15 minutes, followed by another EGG recording 5 minutes after eating. Recording continues for 30 minutes, with a sampling frequency of 4Hz.
Gastric electrogastrography (EGG) testing | up to 4 weeks
  The Hefei Scientific Experimental Instrument Factory's GAP-24A high-resolution gastrointestinal electrogastrography analysis system is used for testing. In the fasted state, the subject lies in a supine position, and electrodes are placed on the upper abdomen at the first lead of the gastric antrum (2-4 cm to the right of the midpoint between the xiphoid process and umbilicus) and the second lead of the gastric body (3-5 cm to the left of the midpoint between the xiphoid process and umbilicus, 1 cm upward). Conductive gel is applied locally to the skin, and a baseline EGG recording is made before conducting gastric EGG evaluation. After recording for 30 minutes, subjects are given a standard meal (50% carbohydrates, 25% protein, 25% fat, total energy intake of 570kcal, and 150mL water), which they eat within 15 minutes, followed by another EGG recording 5 minutes after eating. Recording continues for 30 minutes, with a sampling frequency of 4Hz.

SECONDARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) | baseline, pre-intervention
  Evaluate each subject using the GSRS scale
Gastrointestinal Symptom Rating Scale (GSRS) | up to 4 weeks
  Evaluate each subject using the GSRS scale
Gastrointestinal Symptom Rating Scale (GSRS) | up to 8 weeks
  Evaluate each subject using the GSRS scale
Gastrointestinal Symptom Score Questionnaire (GIS) | baseline, pre-intervention
  Evaluate each subject using the GIS scale
Gastrointestinal Symptom Score Questionnaire (GIS) | up to 4 weeks
  Evaluate each subject using the GIS scale
Gastrointestinal Symptom Score Questionnaire (GIS) | up to 8 weeks
  Evaluate each subject using the GIS scale
Nepean Dyspepsia Index (NDI) | baseline, pre-intervention
  Evaluate each subject using the NDI scale
Nepean Dyspepsia Index (NDI) | up to 4 weeks
  Evaluate each subject using the NDI scale
Nepean Dyspepsia Index (NDI) | up to 8 weeks
  Evaluate each subject using the NDI scale
Functional Dyspepsia Quality of Life questionnaire (FDQOL). | baseline, pre-intervention
  Evaluate each subject using the FDQOL scale
Functional Dyspepsia Quality of Life questionnaire (FDQOL). | up to 4 weeks
  Evaluate each subject using the FDQOL scale
Functional Dyspepsia Quality of Life questionnaire (FDQOL). | up to 8 weeks
  Evaluate each subject using the FDQOL scale
Gastrointestinal hormone level testing | baseline, pre-intervention
  5mL of venous blood is drawn from the subject in a fasted state. After centrifugation at 3000 rpm for 10 minutes at 4℃, the plasma is separated and stored in a -80℃freezer. ELISA method is used to test the levels of MTL, Ghrelin, 5-HT, CCK, PYY, and GLP-1.
Gastrointestinal hormone level testing | up to 4 weeks
  5mL of venous blood is drawn from the subject in a fasted state. After centrifugation at 3000 rpm for 10 minutes at 4℃, the plasma is separated and stored in a -80℃freezer. ELISA method is used to test the levels of MTL, Ghrelin, 5-HT, CCK, PYY, and GLP-1.
Intestinal microbiota diversity testing | baseline, pre-intervention
  Approximately 5g of feces are collected using a sterile fecal collection tube from each subject anytime within three days before and after the start of intervention. The central portion of the feces is collected to avoid contamination with urine or other substances. Diarrhea or loose stools are excluded. The feces samples are stored in a -80℃ freezer for measurement. The QIAamp Fast DNA Stool kit is used for fecal DNA extraction, and 16S rDNA sequencing technology is used to analyze the composition and diversity of the intestinal microbial communities.
Intestinal microbiota diversity testing | up to 4 weeks
  Approximately 5g of feces are collected using a sterile fecal collection tube from each subject anytime within three days before and after the start of intervention. The central portion of the feces is collected to avoid contamination with urine or other substances. Diarrhea or loose stools are excluded. The feces samples are stored in a -80℃ freezer for measurement. The QIAamp Fast DNA Stool kit is used for fecal DNA extraction, and 16S rDNA sequencing technology is used to analyze the composition and diversity of the intestinal microbial communities.
Intestinal microbiota metabolite testing | baseline, pre-intervention
  Non-targeted metabolomics detection method is used to measure the content of SCFAs before and after intervention in healthy volunteers and each group using chromatography-mass spectrometry technology.
Intestinal microbiota metabolite testing | up to 4 weeks
  Non-targeted metabolomics detection method is used to measure the content of SCFAs before and after intervention in healthy volunteers and each group using chromatography-mass spectrometry technology.

IPD SHARING:
Plan to Share IPD: No